CLINICAL TRIAL: NCT06561672
Title: Paracetamol Plus Tramadol Versus Fentanyl As Preemptive Analgesia For Enhanced Recovery
Brief Title: Paracetamol Plus Tramadol Versus Fentanyl As Preemptive Analgesia For Enhanced Recovery After Day Case Surgeries
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Mohamed Medhat, assistant professor of anesthesia and surgical intensive care(Principal Investigator), Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 459
Record Dates: First submitted 2024-08-15; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Preemptive Paracetamol Plus Tramadol and Preemptive Fentanyl
Keywords: paracetamol ,tramadol , fentanyl, day case surgeries
MeSH Terms: interventions — Tramadol; Acetaminophen; Fentanyl; Propofol; cisatracurium

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tramadol plus paracetamol (T) (Experimental)
  Interventions: Drug: tramadol plus paracetamol; Drug: propofol and muscle relaxant (cisatracurium)
- fentanyl(F) (Experimental)
  Interventions: Drug: Fentanyl; Drug: Propofol

INTERVENTIONS:
Drug: tramadol plus paracetamol — Intravenous infusion of 15mg/kg paracetamol together with 1mg/kg tramadol will be started and to be finished before starting of induction of anesthesia (induction agent will be propofol 2mg/kg and muscle relaxant (cisatracurium) 0.15 mg/kg)
  Arms: tramadol plus paracetamol (T)
Drug: Fentanyl — Intravenous injection of 1.5 microgram/kg fentanyl will be given to the patient followed by induction agents (propofol 2mg/kg).
  Arms: fentanyl(F)
Drug: propofol and muscle relaxant (cisatracurium) — propofol 2mg/kg and muscle relaxant (cisatracurium) 0.15 mg/kg)
  Arms: tramadol plus paracetamol (T)
Drug: Propofol — propofol 2mg/kg
  Arms: fentanyl(F)

SUMMARY:
Implementation of enhanced recovery in day case surgeries using either preemptive intravenous paracetamol plus tramadol or preemptive intravenous fentanyl.

DETAILED DESCRIPTION:
after being informed about the study and potential risks. All patients giving written consent will be randomized by double blind manner into two equal groups (T group and F group). Using computer generated randomization table; each group consists of 51 patients:Group (T) (n=51): Patients will receive preemptive intravenous infusion of tramadol plus paracetamol .

Group (F) (n=51): Patients will receive preemptive intravenous fentanyl.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for day case surgeries.
* Patient acceptance to be included into the study.
* Both sex.
* Patients with ASA physical status I, II.
* BMI 25 - 30 kg m-2.
* Duration of surgery from 1-2 hours

Exclusion Criteria:

-Uncooperative patients and patients with psychological problems.-

* Patients with liver or renal impairment.
* Patients with history of allergy to drug used in the study.
* Patients with chronic pain.
* Patient on pain therapy.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Enhanced recovery score | at the end of 24 hour after surgery.
  A 40-item questionnaire that provides a score (QoR-40) that measure quality of recovery after surgery and anesthesia (enhanced recovery) according to five aspects will be recorded at the end of 24 hours after surgery: Emotional state(n=9) physical comfort(n=12) Psychological support (n=7) physical independence(n=5) pain(n=7)
  - Each one of the 40 questions gets a score from one to five at which one is the worst response and five is the best response. When the individual score of all questions are added together we get a total score that ranges from 40 to 200.

SECONDARY OUTCOMES:
The duration of PACU stay | 2 days postoperative
  time from patient admission to the PACU till discharge from the PACU
Duration of postoperative hospital stay | 2 days postoperative
  time from patient admission to the PACU till the hospital discharge admission to the PACU till the hospital discharge
Postoperative pain severity | recorded upon arrival to recovery room and at 1, 2, 4, 6 and 12hours postoperatively based
  (a 10-cm line labeled with "worst pain imaginable" on the right border and "no pain" on the left border).
postoperative agitation score | immediately after extubation, on arrival to PACU, 10 minutes and 20 minutes after arrival to PACU:
  Score Term Description
  * 4 Combative Overtly combative, violent, immediate danger to staff
  * 3 Very agitated Pulls or removes tubes (s) or catheter(s); aggressive
  * 2 Agitated Frequent non-purposeful movement
  * 1 Restless Anxious, but not aggressive or vigorous 0 Alert and calm
    * 1 Drowsy Not fully alert but has sustained awakening (eye opening or eye contact) to voice (< 10 seconds)
    * 2 Light sedation Briefly awaken with eye contact to voice (> 10 seconds)
    * 3 Moderate sedation Movement or eye opening to voice (but no eye contact)-4 Deep sedation No response to voice, but movement or eye opening to physical stimulation
    * 5 Unarousable No response to voice or physical stimulation

CONTACTS AND LOCATIONS:
Overall Officials: marwa M Medhat, MD, Principal Investigator — Zagazig University
Locations (1):
- Aculty of Medicine,Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No